CLINICAL TRIAL: NCT03783975
Title: A Community-Based Approach to Overcoming Barriers to Cascade Screening for Long QT Syndrome
Brief Title: KCNQ1 Cascade Screening
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain all survey data due to COVID delay
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Amber Beitelshees, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HP-00081981; R21HG010412 (NIH)
Record Dates: First submitted 2018-12-18; First posted 2018-12-21 (Actual); Results first posted 2022-10-26 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Long QT Syndrome
Keywords: Cascade; Screening; Ethical; Legal; Social
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simplified Cascade Screening (Experimental): Free, mail-in, saliva-based screening for the KCNQ1 Thr224Met variant.
  Interventions: Genetic: Simplified Cascade Screening

INTERVENTIONS:
Genetic: Simplified Cascade Screening — Screening of the KCNQ1 Thr224Met variant for family members of probands

SUMMARY:
The objectives of the protocol are to: (1) evaluate the uptake of cascade screening and preventative therapies after the implementation of a simplified screening process and (2) assess proband and family member perspectives about the return of research results and cascade screening for the KCNQ1 Thr224Met variant. The investigators will conduct a mixed methods study in the Old Order Amish community where the KCNQ1 variant is enriched over 100,000-fold compared to other populations. The intervention will offer free, mail-in, saliva-based genetic testing for family members of probands. The rate of uptake of testing and preventative therapy after the intervention is implemented (i.e. when 'simplified' free, mail-in, saliva-based testing was available) will be compared to data from before the intervention (i.e. when 'traditional' $50 blood-based testing was available to family members) when uptake was essentially zero. The primary outcome is the rate of uptake of cascade screening with the intervention ('simplified'). The secondary outcomes include: extent of disclosure of genotype results before and after the intervention, proportion of informed relatives who get screened before and after the intervention, and the uptake of appropriate preventative care (e.g. seeing a cardiologist and/or taking beta-blocker). The tertiary outcomes are demographic characteristics associated with uptake of cascade screening or uptake of preventative therapy. The investigators will also assess qualitative themes surrounding the return of results process and cascade screening using interviews.

ELIGIBILITY:
Inclusion Criteria:

* KCNQ1Thr224Met proband or first degree family member

Exclusion Criteria:

* Family members who have not been contacted by probands

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 131 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2022-12-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Amish Research Clinic, Lancaster, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Simplified Cascade Screening
Started | 131
Completed | 131
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Simplified Cascade Screening
Number analyzed (Participants) | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 88
  Between 18 and 65 years | 41
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 131
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 131

OUTCOME MEASURES:

1. Primary Outcome: Percentage of At-risk Family Members Who Underwent Cascade Screening
Description: Rate of uptake of cascade screening after the intervention ('simplified')
Time Frame: 18 months
Population: 809 family members were eligible to be screened and were considered at-risk.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplified Cascade Screening
Number analyzed (Participants) | 809
Participants | 131

2. Secondary Outcome: Extent of Disclosure Determined by Questionnaire
Description: proportion of family members told after the intervention ('simplified')
Time Frame: 18 months
Population: Because of COVID, too much time had passed since we had originally contacted the probands and we did not think we could get reliable data on how many family members they had told after the intervention. Thus, these data were not collected. During the COVID pandemic we had to switch gears and warn people with LQTS about the risks of QT-prolongation with chloroquine, hydroxychloroquine, and azithromycin.
Arm/Group | Simplified Cascade Screening
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Informed Relatives Screened Determined by Questionnaire
Description: Number of informed family members tested after the intervention ('simplified')
Time Frame: 18 months
Population: Number of family members tested of those mailed letters. The overall number of participants analyzed differs from the number in the Participant Flow Module because it represents the number of family members who were mailed letters whereas the participant flow module includes individuals who consented for testing. These numbers are not related to each other because we didn't mail letters to children, although children were eligible for testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplified Cascade Screening
Number analyzed (Participants) | 145
Participants | 27

4. Secondary Outcome: Number of Participants With an Uptake of Preventative Therapy as Determined by Questionnaire
Description: Uptake of preventative therapy was defined as those taking a beta-blocker if recommended or those who implemented lifestyle modifications if beta-blocker not recommended. The survey was mailed to all probands.
Time Frame: 18 months
Population: We analyzed the number of survey responses obtained for the questions on beta-blocker therapy and lifestyle modifications which is why the numbers are different than those reported in the participant flow module.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplified Cascade Screening
Number analyzed (Participants) | 31
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse events were obtained at the time of saliva sample collection.
Description: Adverse events were obtained at the time of enrollment when saliva samples were collected. All other study procedures were surveys.
Arm/Group | Simplified Cascade Screening
All-Cause Mortality (participants affected / at risk) | 0/131
Serious Adverse Events (participants affected / at risk) | 0/131
Other Adverse Events (participants affected / at risk) | 0/131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT03783975/Prot_SAP_000.pdf